CLINICAL TRIAL: NCT00567203
Title: A Phase 1B Inpatient, Randomized, Double-Blind, Placebo-Controlled, Crossover Study Of The Safety And Efficacy Of Two Fixed Doses Of PF-3463275 In Adjunctive Treatment Of Cognitive Deficits In Schizophrenia
Brief Title: A Study Of Adjunctive Treatment Of Cognitive Deficits In Schizophrenia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trials Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: A9131004
Record Dates: First submitted 2007-12-03; First posted 2007-12-04 (Estimated); Last update posted 2008-10-02 (Estimated); Status verified 2008-10

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — 1-methyl-1H-imidazole-4-carboxylic acid (3-chloro-4-fluoro-benzyl)-(3-methyl-3-aza-bicyclo(3.1.0) hex-6-ylmethyl)amide

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental)
  Interventions: Drug: PF-3463275
- 2 (Experimental)
  Interventions: Drug: PF-3463275
- 3 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PF-3463275 — PF-3463275 10mg
  Arms: 1
Drug: PF-3463275 — PF-3463275 25mg
  Arms: 2
Drug: Placebo — Placebo
  Arms: 3

SUMMARY:
The objective of this study is to evaluate the safety, tolerability, and efficacy of two dose regimens of PF-3463275 compared with placebo added to ongoing atypical antipsychotic therapy for cognitive deficits in subjects with chronic symptoms of schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of schizophrenia
* In stable treatment with risperidone, olanzapine, quetiapine, ziprasidone, aripiprazole, or paliperidone for at least 2 months
* Stable symptoms of schizophrenia for at least 3 months.

Exclusion Criteria:

* Subjects with a psychiatric disorder other than schizophrenia
* Substance dependence or abuse
* Women who have child bearing potential.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2007-11; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the CNS Vital Signs Cognition Battery composite score | 6 days
Safety Endpoints: tolerability, laboratory tests, vital signs, and ECG's. | 38 days
Pharmacokinetics of PF-3463275 | 6 days

SECONDARY OUTCOMES:
Positive and Negative Syndrome Scale (PANSS) | 6 days
Change from baseline in the CNS Vital Signs Cognition Battery domain scores | 6 days

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- United States (2):
  - Pfizer Investigational Site, Glendale, California
  - Pfizer Investigational Site, Willingboro, New Jersey

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A9131004&StudyName=A%20Study%20Of%20Adjunctive%20Treatment%20Of%20Cognitive%20Deficits%20In%20Schizophrenia